CLINICAL TRIAL: NCT03167801
Title: Melatonin Secretion and Sleep Quality in Spinal Cord Injury Patients
Acronym: MELATETRA
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A00605-46
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Spinal Cord Injuries
Keywords: tetraplegia; spinal cord injury; melatonin; sleep quality; sleepiness
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Sleep Initiation and Maintenance Disorders; Sleepiness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spinal cord injury: spinal cord injury all scores AIS
- Healthy volunteers: Healthy volunteers for whom melatonin profiles have been taken and stored in the Lyon endocrinology laboratory's database. No healthy volunteers will be directly recruited for the study.

SUMMARY:
To evaluate the relationship between secretion of melatonin and sleep quality in spinal cord injury patients versus a database of healthy volunteers.

DETAILED DESCRIPTION:
Melatonin is a neurohormone secreted by the pineal gland and excreted by the urinary tract. It has a key role in the synchronisation of circadian rhythms including the sleep wake cycle, with a peak secretion around 03:00.

The neural pathway controlling melatonin secretion is long and transits via the thoracic spine. The exact level is not known, but interruption of the connection in patients with lesions of the spinal cord is known to occur.

Tetraplegic patients often complain of insomnia, daytime sleepiness and poor sleep quality but the contribution of melatonin levels to sleep quality has not been explored in large studies, although case reports have shown reduced or abolished melatonin secretion and altered melatonin secretion profiles with delayed peak secretion. Paraplegic patients report fewer sleep difficulties and little is known about melatonin secretion in this group. The investigators hypothesize that sleep abnormalities are related to abnormalities in melatonin secretion and that this is in turn related to the level of the spinal cord injury

The study aims to explore the profiles of melatonin secretion in patients with spinal cord injuries and comparing melatonin profiles with a database of healthy volunteers. The investigators will further analyse the results looking at the severity of spinal cord injury using the Abbreviated Injury Scale (AIS) and the level of the injury. Outcome measures are melatonin secretion profile, sleep complaints measured using the Pittsburgh scale and daytime sleepiness measured using the Epworth sleep scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Spinal cord injury patient
* All score AIS
* With a chronic lesion (more than 6 months from initial injury)
* Signed informed consent

Exclusion Criteria:

* Pregnant women
* Breast feeding women
* Refusal to participate at study
* Not covered by national health insurance scheme
* Patient unable to give informed consent
* Transmeridian flight crossing more than 3 time zones in the month preceding the study
* Recent treatment with melatonin (< 1 month) or beta blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal cord injury patients
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Urinary 6-sulfatoxy-melatonin (U6SM) | 24 hours
  Urinary 6-sulfatoxy-melatonin (U6SM) will be measured during 24 hours

SECONDARY OUTCOMES:
Sleep quality | 24 hours
  Pittsburgh Sleep Quality Index
Daytime sleepiness | 24 hours
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonia Quera-Salva, MD-PhD, Study Director — APHP Hopital Raymond Poincare; Raphaella Daville, MD, Principal Investigator — APHP Hopital Raymond Poincare; Djamel BENSMAIL, MD-PhD, Study Chair — APHP Hopital Raymond Poincare
Locations (1):
- APHP Hôpital Raymond poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No